CLINICAL TRIAL: NCT01571414
Title: A Phase I, Three-Arm Safety, Tolerability, and Pharmacokinetic Interaction Study of PA-824, an Investigational Nitroimidazole for the Treatment of Tuberculosis, Together With Efavirenz, Ritonavir-Boosted Lopinavir, or Rifampin
Brief Title: Evaluating the Safety and Drug Interaction of PA-824, an Investigational Tuberculosis Medication, Together With Efavirenz, Ritonavir-Boosted Lopinavir, or Rifampin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A5306; 11829 (Registry Identifier: DAIDS ES Registry Number); ACTG5306
Record Dates: First submitted 2012-03-20; First posted 2012-04-05 (Estimated); Last update posted 2021-11-05 (Actual); Status verified 2015-04

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — pretomanid; efavirenz; Lopinavir; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Arm 1A-EFV and PA-824 (Experimental): Participants will receive PA-824 on Days 1 to 7, no study medication on Days 8 to 21, EFV on Days 22 to 35, and EFV plus PA-824 on Days 36 to 42. Inpatient study visits will occur at Days 7, 34, and 41 to 42.
  Interventions: Drug: PA-824; Drug: Efavirenz (EFV)
- Arm 1B-EFV and PA-824 (Experimental): Participants will receive EFV on Days 1 to 14, EFV plus PA-824 on Days 15 to 21, no study medication on Days 22 to 35, and PA-824 on Days 36 to 42. Inpatient study visits will occur at Days 13, 20 to 21, and 42.
  Interventions: Drug: PA-824; Drug: Efavirenz (EFV)
- Arm 2A-LPV/r and PA-824 (Experimental): Participants will receive PA-824 on Days 1 to 7, no study medication on Days 8 to 21, LPV/r on Days 22 to 35, and LPV/r plus PA-824 on Days 36 to 42. Inpatient study visits will occur at Days 7, 35, and 42.
  Interventions: Drug: PA-824; Drug: Lopinavir/Ritonavir (LPV/r)
- Arm 2B-LPV/r and PA-824 (Experimental): Participants will receive LPV/r on Days 1 to 14, LPV/r plus PA-824 on Days 15 to 21, no study medication on Days 22 to 35, and PA-824 on Days 36 to 42. Inpatient study visits will occur at Days 14, 21, and 42.
  Interventions: Drug: PA-824; Drug: Lopinavir/Ritonavir (LPV/r)
- Arm 3-RIF and PA-824 (Experimental): Participants will receive PA-824 on Days 1 to 7, RIF on Days 8 to 14, and RIF plus PA-824 on Days 15 to 21. Inpatient study visits will occur at Days 7 and 21.
  Interventions: Drug: PA-824; Drug: Rifampin (RIF)

INTERVENTIONS:
Drug: PA-824 — 200-mg tablets once a day
Drug: Efavirenz (EFV) — 600-mg tablets once a day
  Arms: Arm 1A-EFV and PA-824; Arm 1B-EFV and PA-824
Drug: Lopinavir/Ritonavir (LPV/r) — 400-mg/100-mg tablets twice a day
  Arms: Arm 2A-LPV/r and PA-824; Arm 2B-LPV/r and PA-824
Drug: Rifampin (RIF) — 300-mg capsules once a day
  Arms: Arm 3-RIF and PA-824

SUMMARY:
Tuberculosis (TB) is a global public health concern and developing new treatment regimens is an important research priority. PA-824 is an experimental TB medication. This study will evaluate the safety and tolerability of PA-824 when combined with efavirenz (EFV) or ritonavir-boosted lopinavir (LPV/r), which are medications used to treat HIV infection, or rifampin (RIF), which is a medication used to treat TB. Study researchers will examine the safety and tolerability of these drug combinations and how the medications affect the levels of PA-824 in the blood.

DETAILED DESCRIPTION:
TB is a global public health threat. In 2009, there were an estimated 9.4 million cases of TB and 1.8 million deaths from the disease. TB treatment regimens are often lengthy and complex, and multidrug-resistant (MDR) TB is emerging as a worldwide epidemic. TB is also one of the most common causes of death among people infected with HIV. PA-824 is an experimental drug developed for the treatment of TB. This study will evaluate the safety, tolerability, and pharmacokinetic (PK) drug interactions between PA-824 and EFV, LPV/r, or RIF.

This study will enroll healthy adults who are not infected with HIV or TB. Participants will be enrolled into one of three arms, with Arms 1 and 2 each consisting of two groups. Participants in Arm 1 will be randomly assigned to receive PA-824 alone or EFV alone followed by EFV plus PA-824 in one of two sequences. Participants in Arm 2 will be randomly assigned to receive PA-824 alone or LPV/r alone followed by LPV/r plus PA-824 in one of two sequences. For participants in Arms 1 and 2, there will be a 14-day washout period between treatments, where participants will not receive any medication. Participants in Arm 3 will receive PA-824 alone, followed by RIF alone, and then RIF plus PA-824. Participants in Arms 1 and 2 will attend outpatient study visits at study entry and either Days 3, 22, and 29 or Days 7, 36, and 39, depending on which group they are in. Participants in Arm 3 will attend outpatient study visits at study entry and Days 3, 10, and 15. At most study visits, participants will undergo a physical examination, vital sign measurements, medication and medical history review, and blood collection. Participants will complete a medication and symptom diary throughout the study.

All participants also will be admitted to an inpatient clinical research unit two or three times during the study, depending on which arm they are enrolled in. Each inpatient visit will last 1 or 2 days. During the inpatient visits, participants will undergo several blood collections throughout the day; select visits also will include an electrocardiogram (ECG).

Participants in Arms 1 and 2 will receive the last dose of their assigned medication on Day 42. Participants in Arm 3 will receive the last dose of their assigned medication on Day 21. A final study visit will occur for all participants 1 to 2 weeks later.

ELIGIBILITY:
Inclusion Criteria:

* Contraception requirements: Females of reproductive potential must have a negative serum or urine beta-human choriogonadotropin (β-HCG) pregnancy test performed within 48 hours before study entry. All participants must agree not to participate in a conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization). If participating in sexual activity that could lead to pregnancy, participants must agree to use two reliable forms of contraceptives simultaneously while on study and for a number of weeks after the final study visit as defined in the protocol. More information on this criterion can be found in the protocol.
* Able and willing to provide written informed consent
* Absence of HIV-1 infection, as documented by any licensed enzyme-linked immunosorbent assay (ELISA) test kit, within 21 days prior to study entry
* Creatinine clearance of greater than 50 mL/min, within 21 days prior to study entry, calculated by the Cockcroft-Gault method. More information on this criterion can be found in the protocol.
* Laboratory values obtained within 21 days prior to study entry:

  1. Hemoglobin greater than 12 g/dL for men and greater than 11 g/dL for women
  2. Platelet count greater than or equal to 125,000/cu mm
  3. Absolute neutrophil count greater than or equal to 1,250/cu mm
  4. Serum albumin greater than or equal to the lower limit of normal for the laboratory
  5. Serum potassium greater than or equal to the lower limit of normal and less than or equal to the upper limit of normal for the laboratory
  6. Serum alanine aminotransferase (ALT) less than or equal to the upper limit of normal (ULN) for the laboratory
* Note: Screening laboratory evaluations may be repeated if one or more of the values are out of range. It is preferable, although not required, for prospective participants to fast (i.e., nothing by mouth [NPO] except water) for 4 hours prior to drawing samples for screening serum albumin, serum potassium, and serum ALT evaluations.
* Hepatitis B surface antigen negative, performed by a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory within 21 days prior to study entry
* Hepatitis C virus (HCV) antibody negative or, if the participant is known to have a positive hepatitis C antibody test, negative HCV RNA test, performed by a CLIA-certified laboratory within 21 days prior to study entry

Exclusion Criteria:

* Use of any prescription or nonprescription medication known to inhibit or induce CYP3A or CYP2B6 metabolizing enzymes (refer to the manufacturers' package inserts for individual drugs) within 30 days prior to study entry
* Planned use during the study, from study entry through the last PK blood draw, of any of the following: prescription medication(s) [excluding IUDs that elute locally active hormonal contraceptives], herbal supplement(s), nutritional supplement(s), or over-the-counter medication(s). Note: Multivitamins, acetaminophen (up to 650 mg every 6 hours as an analgesic), ibuprofen (up to 600 mg twice daily), naproxen (up to 500 mg twice daily for pain or headache), and diphenhydramine (up to 25 mg daily for insomnia or seasonal allergies) are permitted.
* Hospitalization for any reason within 14 days prior to study entry
* Pharmacotherapy for serious illness within 14 days prior to study entry
* Use of any prescription medication(s) within 14 days prior to study entry
* Receipt of any investigational study drug, vaccine, or treatment within 21 days prior to study entry
* Known allergy/sensitivity or any hypersensitivity to PA-824, EFV, LPV, RTV, RIF, or components of their formulations
* As determined by the site investigator, a significant previous or active history of cardiovascular, renal, liver, hematologic, neurologic, gastrointestinal, psychiatric, endocrine, or immunologic disease(s); this is inclusive of chronic illnesses or gastrointestinal conditions that may affect drug absorption, etc.
* Any medical condition that, in the opinion of the site investigator, would interfere with the participant's ability to participate in the study
* Active illicit drug use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Clinical evidence of active TB. Note: Clinical evidence of active TB is based on history and physical examination. No other screening tests for TB are required for the study.
* Inability to abstain from consuming alcoholic beverages during defined periods throughout the study and grapefruits, mandarin oranges, and grapefruit juice for the entire duration of the study. Note: Participants are permitted to consume alcoholic beverages only during the washout period of Arms 1 and 2. Participants must agree to abstain from consuming alcoholic beverages for the duration of Arm 3.
* For smokers, inability to smoke less than or equal to 5 cigarettes per day for the entire duration of the study
* Breastfeeding
* ECG showing first-degree or greater heart block or QTc greater than 450 ms within 21 days prior to study entry. More information on this criterion can be found in the protocol.
* Frequent or severe headaches, defined as more than two headaches per week on average during the last 30 to 60 days prior to study entry or headaches greater than or equal to once every 30 days during the last 90 days prior to study entry that were severe enough to interfere with activities of daily living or ability to work or carry out daily responsibilities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Arm 1: PA-824 PK parameters area under the concentration-time curve (AUC) of 24 hours when dosed alone and when dosed together with EFV 600 mg daily | Measured at participants' inpatient study visits at Days 7, 34, and 41 to 42 (Arm 1A) and at Days 13, 20 to 21, and 42 (Arm 1B)
Arm 1: Grade 2 or higher signs and symptoms observed while on study and during the follow-up | Measured through participants' last study visit at Days 49 to 56
Arm 2: PA-824 PK parameters AUC of 24 hours when dosed alone and when dosed together with LPV/r 400/100 mg twice daily | Measured at participants' inpatient study visits at Days 7, 35, and 42 (Arm 2A) and at Days 14, 21, and 42 (Arm 2B)
Arm 2: Grade 2 or higher signs and symptoms observed while on study and during the follow-up | Measured through participants' last study visit at Days 49 to 56
Arm 3: PA-824 PK parameters AUC of 24 hours when dosed alone and when dosed together with RIF 600 mg once daily | Measured at participants' inpatient study visits at Days 7 and 21
Arm 3: Grade 2 or higher signs and symptoms observed while on study and during the follow-up | Measured through participants' last study visit at Days 29 to 36
Arm 1: PA-824 PK parameters Cmax when dosed alone and when dosed together with EFV 600 mg daily | Measured at participants' inpatient study visits at Days 7, 34, and 41 to 42 (Arm 1A) and at Days 13, 20 to 21, and 42 (Arm 1B)
Arm 2: PA-824 PK parameters Cmax when dosed alone and when dosed together with LPV/r 400/100 mg twice daily | Measured at participants' inpatient study visits at Days 7, 35, and 42 (Arm 2A) and at Days 14, 21, and 42 (Arm 2B)
Arm 3: PA-824 PK parameters Cmax when dosed alone and when dosed together with RIF 600 mg once daily | Measured at participants' inpatient study visits at Days 7 and 21

SECONDARY OUTCOMES:
Arm 1: PA-824 PK parameters Cmin when dosed alone and when dosed together with EFV 600 mg daily | Measured at participants' inpatient study visits at Days 7, 34, and 41 to 42 (Arm 1A) and at Days 13, 20 to 21, and 42 (Arm 1B)
Arm 1: EFV PK parameters AUC of 24 hours when EFV is dosed alone and when dosed together with PA-824 200 mg daily | Measured at participants' inpatient study visits at Days 7, 34, and 41 to 42 (Arm 1A) and at Days 13, 20 to 21, and 42 (Arm 1B)
Arm 2: PA-824 PK parameters Cmin when dosed alone and when dosed together with LPV/r 400/100 mg twice daily | Measured at participants' inpatient study visits at Days 7, 35, and 42 (Arm 2A) and at Days 14, 21, and 42 (Arm 2B)
Arm 2: LPV PK parameters AUC of 12 hours when LPV/r is dosed alone and when dosed together with PA-824 200 mg daily | Measured at participants' inpatient study visits at Days 7, 35, and 42 (Arm 2A) and at Days 14, 21, and 42 (Arm 2B)
Arm 3: PA-824 PK parameters Cmin when dosed alone and when dosed together with RIF 600 mg daily | Measured through participants' last study visit at Days 29 to 36
Arm 1: PA-824 PK parameters T1/2 when dosed alone and when dosed together with EFV 600 mg daily | Measured at participants' inpatient study visits at Days 7, 34, and 41 to 42 (Arm 1A) and at Days 13, 20 to 21, and 42 (Arm 1B)
Arm 1: PA-824 PK parameters CL/F when dosed alone and when dosed together with EFV 600 mg daily | Measured at participants' inpatient study visits at Days 7, 34, and 41 to 42 (Arm 1A) and at Days 13, 20 to 21, and 42 (Arm 1B)
Arm 1: EFV PK parameters Cmax when EFV is dosed alone and when dosed together with PA-824 200 mg daily | Measured at participants' inpatient study visits at Days 7, 34, and 41 to 42 (Arm 1A) and at Days 13, 20 to 21, and 42 (Arm 1B)
Arm 1: EFV PK parameters Cmin when EFV is dosed alone and when dosed together with PA-824 200 mg daily | Measured at participants' inpatient study visits at Days 7, 34, and 41 to 42 (Arm 1A) and at Days 13, 20 to 21, and 42 (Arm 1B)
Arm 1: EFV PK parameters CL/F when EFV is dosed alone and when dosed together with PA-824 200 mg daily | Measured at participants' inpatient study visits at Days 7, 34, and 41 to 42 (Arm 1A) and at Days 13, 20 to 21, and 42 (Arm 1B)
Arm 1: EFV PK parameters T1/2 when EFV is dosed alone and when dosed together with PA-824 200 mg daily | Measured at participants' inpatient study visits at Days 7, 34, and 41 to 42 (Arm 1A) and at Days 13, 20 to 21, and 42 (Arm 1B)
Arm 2: PA-824 PK parameters T1/2 when dosed alone and when dosed together with LPV/r 400/100 mg twice daily | Measured at participants' inpatient study visits at Days 7, 35, and 42 (Arm 2A) and at Days 14, 21, and 42 (Arm 2B)
Arm 2: PA-824 PK parameters CL/F when dosed alone and when dosed together with LPV/r 400/100 mg twice daily | Measured at participants' inpatient study visits at Days 7, 35, and 42 (Arm 2A) and at Days 14, 21, and 42 (Arm 2B)
Arm 2: LPV PK parameters Cmax when LPV/r is dosed alone and when dosed together with PA-824 200 mg daily | Measured at participants' inpatient study visits at Days 7, 35, and 42 (Arm 2A) and at Days 14, 21, and 42 (Arm 2B)
Arm 2: LPV PK parameters Cmin when LPV/r is dosed alone and when dosed together with PA-824 200 mg daily | Measured at participants' inpatient study visits at Days 7, 35, and 42 (Arm 2A) and at Days 14, 21, and 42 (Arm 2B)
Arm 2: LPV PK parameters CL/F when LPV/r is dosed alone and when dosed together with PA-824 200 mg daily | Measured at participants' inpatient study visits at Days 7, 35, and 42 (Arm 2A) and at Days 14, 21, and 42 (Arm 2B)
Arm 2: LPV PK parameters T1/2 when LPV/r is dosed alone and when dosed together with PA-824 200 mg daily | Measured at participants' inpatient study visits at Days 7, 35, and 42 (Arm 2A) and at Days 14, 21, and 42 (Arm 2B)
Arm 3: PA-824 PK parameters T1/2 when dosed alone and when dosed together with RIF 600 mg daily | Measured at participants' inpatient study visits at Days 7 and 21
Arm 3: PA-824 PK parameters CL/F when dosed alone and when dosed together with RIF 600 mg daily | Measured at participants' inpatient study visits at Days 7 and 21

CONTACTS AND LOCATIONS:
Overall Officials: Kelly E. Dooley, MD, PhD, Study Chair — Johns Hopkins University
Locations (4):
- United States (4):
  - Ucsf Hiv/Aids Crs, San Francisco, California
  - Johns Hopkins University CRS, Baltimore, Maryland
  - Ohio State University CRS, Columbus, Ohio
  - Vanderbilt Therapeutics (VT) CRS, Nashville, Tennessee

REFERENCES:
- [Background] Lenaerts AJ, Gruppo V, Marietta KS, Johnson CM, Driscoll DK, Tompkins NM, Rose JD, Reynolds RC, Orme IM. Preclinical testing of the nitroimidazopyran PA-824 for activity against Mycobacterium tuberculosis in a series of in vitro and in vivo models. Antimicrob Agents Chemother. 2005 Jun;49(6):2294-301. doi: 10.1128/AAC.49.6.2294-2301.2005. PMID 15917524
- [Background] Singh R, Manjunatha U, Boshoff HI, Ha YH, Niyomrattanakit P, Ledwidge R, Dowd CS, Lee IY, Kim P, Zhang L, Kang S, Keller TH, Jiricek J, Barry CE 3rd. PA-824 kills nonreplicating Mycobacterium tuberculosis by intracellular NO release. Science. 2008 Nov 28;322(5906):1392-5. doi: 10.1126/science.1164571. PMID 19039139
- [Derived] Dooley KE, Luetkemeyer AF, Park JG, Allen R, Cramer Y, Murray S, Sutherland D, Aweeka F, Koletar SL, Marzan F, Bao J, Savic R, Haas DW; AIDS Clinical Trials Group A5306 Study Team. Phase I safety, pharmacokinetics, and pharmacogenetics study of the antituberculosis drug PA-824 with concomitant lopinavir-ritonavir, efavirenz, or rifampin. Antimicrob Agents Chemother. 2014 Sep;58(9):5245-52. doi: 10.1128/AAC.03332-14. Epub 2014 Jun 23. PMID 24957823